CLINICAL TRIAL: NCT03857360
Title: Effectiveness of PENTABIOCEL in Clinical and Laboratory Recovery of Children With Celiac Disease: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Effectiveness of PENTABIOCEL in Clinical and Laboratory Recovery of Children With Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Noos S.r.l. (Industry)
Responsible Party: Principal Investigator, Carlo Catassi, M.D., Professor and Head, Department of Pediatrics, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CD-PENTABIOCEL
Record Dates: First submitted 2019-02-13; First posted 2019-02-28 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Celiac Disease
Keywords: Gluten; Probiotic; Microbiota; Dysbiosis
MeSH Terms: conditions — Celiac Disease; Dysbiosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentabiocel (Active Comparator): Oral administration of one sachet of Pentabiocel for 12 consecutive weeks.
  Interventions: Dietary Supplement: Pentabiocel
- Placebo (Placebo Comparator): Oral administration of one sachet of Placebo per day for 12 consecutive weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pentabiocel — Pentabiocel is the trade name of the product containing the probiotic mixture of: Lactobacillus paracasei LMG P-17504, Lactobacillus plantarum CECT 4528, Bifidobacterium breve Bbr8 LMG P-17501, Bifidobacterium breve BL10 LMG P-17500 and Bifidobacterium animalis subsp lactis Bi1 LMG P -17,502.
  Arms: Pentabiocel
Dietary Supplement: Placebo — Placebo is composed of maltodextrin which is easily digestible, being absorbed as rapidly as glucose. Maltodextrin listed by the U.S. Food and Drug Administration (FDA) as a safe food additive.
  Arms: Placebo

SUMMARY:
Celiac disease (CD) is an inflammatory condition of the small intestine. Environmental and genetic factors are involved in the development of CD. Apart from environmental and genetic factors other factors may also be involved, such as alteration in intestinal microbiota. Probiotic supplementation has been shown to be able to determine the intestinal healing. Recently the use of a mixture of some specific bacterial strains has shown its effectiveness. In this study effectiveness of a probiotic "Pentabiocel" which is a mixture of five different bacterial strains will be evaluated in CD affected children (already on a gluten-free diet) through a double-blind randomised placebo control trial.

DETAILED DESCRIPTION:
Celiac disease (CD) is an intestinal inflammatory condition characterized by permanent intolerance to gluten, a protein complex present in wheat, barley, and rye, in genetically predisposed subjects. In the early phase of the disease, specific autoantibodies are generally present, which is relevant for diagnostic purposes (especially anti-tissue transglutaminase antibodies (anti TTG) of IgA (immunoglobulin A) class and anti-endomysial antibodies( EMA), and a duodenal and jejunal mucosal lesion that is characterized by an increase in intraepithelial lymphocytes (IEL), hypertrophy of crypts and villous atrophy. The only accepted and effective treatment for CD so far is a lifelong strict gluten-free diet(GFD).

On the clinical level, CD can have an extremely variable expression, from almost silent forms to cases with more or less striking intestinal and extra-intestinal manifestations. Treatment with a strict GFD causes gradual normalisation of the intestinal lesion (generally within 12-24 months). The persistence of a minimal intestinal lesion and of mostly gastro-enteric symptoms, is not rare in adulthood, especially for the difficulty of maintaining a "zero gluten content" diet over time. The "timing" of recovery induced by the GFD is variable from patient to patient and depends on numerous factors such as presentation mode (typical, atypical or silent), the age of onset, adherence to a strict GFD, etc. Among the factors that may condition the normalisation of the clinical picture. According to some recent data, the quantitative and qualitative typology of the intestinal microbiome may have role. Prospective studies in healthy infants who are at risk of developing CD have shown that the Human Leukocyte Antigen (HLA) genotype, together with other environmental factors, influences the composition of the microbiota. In addition, celiac patients have alterations of the intestinal microbiome (dysbiosis) that do not completely normalize even after starting GFD. It has therefore been suggested that CD may favor dysbiosis which in turn negatively influences intestinal mucosal damage and can promote inflammation through the expansion of harmful bacteria and the reduction of beneficial bacteria.

Probiotics are live microorganisms, that when ingested in appropriate quantities, give to the host benefits. Some probiotics may digest gluten and are thus able to reduce their toxicity when used in fermentation processes. For example, a research group (Di Cagno et al.) has shown that bakery products made using a natural yeast with wheat flour fermented by proteases of lactobacilli and mushrooms, can be taken with confidence by celiac patients. This data suggests that the simple administration of a probiotic is capable to provide benefit in patients with CD leading to an improvement also of intestinal symptoms. However, it is clear from the literature that not all probiotic strains possess this characteristic. It has been shown that a mixture of probiotic strains, in particular belonging to the species Lactobacillus paracasei, Lactobacillus plantarum, Bifidobacterium breve, and Bifidobacterium animalis subsp lactis, is able to significantly improve the irritable colon-like gastrointestinal symptoms of patients with CD. Pentabiocel is the trade name of the product containing the above mentioned probiotic mixture: Lactobacillus paracasei (LMG P-17504), Lactobacillus plantarum (CECT 4528), Bifidobacterium breve Bbr8 (LMG P-17501), Bifidobacterium breve (BL10 LMG P-17500) and Bifidobacterium animalis subsp lactis Bi1 (LMG P -17,502).

In this randomized double blind placebo controlled trial study investigators will investigate the effect of "Pentabiocel" on children already on GFD.

The aim of this study is to evaluate the efficacy of "Pentabiocel" in the clinical and laboratory recovery of children with celiac disease

ELIGIBILITY:
Inclusion Criteria:

* Children / adolescents aged between 2 and 16 recruited at the time of diagnosis of celiac disease.

The diagnosis of celiac disease will be performed according to the ESPGHAN 2012 Guidelines.

Exclusion Criteria:

* Patients with autoimmune comorbidity (eg type 1 diabetes) or other associated chronic diseases
* Associated serum IgA selective deficiency
* Poor adherence to gluten free diet at the 6-month control, measured by a score> 10 at the Wessels questionnaire.
* Adherence to the intervention protocol <85%.
* Antibiotic therapy performed during the 7 days preceding T0 and / or T6.
* Antibiotic therapy during the 3 months of probiotic / placebo treatment.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Assessment of recovery time of clinical features | 3 months
  After three months of probiotic treatment patients will be compared with their clinical symptoms evaluating score based Celiac symptom Index (CSI) developed by Leffler DA et al.

SECONDARY OUTCOMES:
Differences between two treatment groups related to all the evaluated parameters | 3 & 6 months
  Differences between the two treatment groups (Placebo and control )related to all the parameters evaluated and in particular: (a) Weight (in kilograms) , height (in meter) will be combined to measure BMI (at the time of enrolment and after follow up 3 and 6 months).
  (b) Anti tissue transglutaminase IgA serology level in cubic inch ( CU) (at the time of enrolment and after follow up 3 and 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Catassi, MPH, Principal Investigator — Univeristà Politecnica delle Marche, Ancona, Italy; Elena Lionett, PhD, Principal Investigator — Univeristà Politecnica delle Marche, Ancona, Italy; Basilio Malamisura, Principal Investigator — Cava de' Tirreni - Ospedale di cava De' tirreni, UO di Pediatria, Salerno, Italy
Locations (1):
- Department of Pediatrics, via Corridoni 11, Ancona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lionetti E, Castellaneta S, Francavilla R, Pulvirenti A, Tonutti E, Amarri S, Barbato M, Barbera C, Barera G, Bellantoni A, Castellano E, Guariso G, Limongelli MG, Pellegrino S, Polloni C, Ughi C, Zuin G, Fasano A, Catassi C; SIGENP (Italian Society of Pediatric Gastroenterology, Hepatology, and Nutrition) Working Group on Weaning and CD Risk. Introduction of gluten, HLA status, and the risk of celiac disease in children. N Engl J Med. 2014 Oct 2;371(14):1295-303. doi: 10.1056/NEJMoa1400697. PMID 25271602
- [Result] Fasano A, Catassi C. Clinical practice. Celiac disease. N Engl J Med. 2012 Dec 20;367(25):2419-26. doi: 10.1056/NEJMcp1113994. No abstract available. PMID 23252527